CLINICAL TRIAL: NCT07329062
Title: Investigation of the Effect of Toothpastes With Different Ingredients on Oral Malodor in Young Adults
Brief Title: Effect of Toothpastes on Oral Malodor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Basak Karasu, Assisstant Professor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Approval No: 18, Date: 29/01/2
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Oral Malodor (Halitosis)
Keywords: Oral Malodor; Propolis; Probiotic toothpaste
MeSH Terms: conditions — Halitosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Propolis containing toothpaste (Experimental): Participants in this arm used propolis containing toothpaste twice daily for routine oral hygiene during the study period.
  Interventions: Other: Propolis Containing Toothpaste
- probiotic containing toothpaste (Experimental): Participants in this arm used probiotic containing toothpaste twice daily for routine oral hygiene during the study period.
  Interventions: Other: Probiotic containing toothpaste
- Phosphate-based formulation toothpaste (Experimental): Participants in this arm used phosphate-based formulation toothpaste twice daily for routine oral hygiene during the study period.
  Interventions: Other: Phosphate-based formulation toothpaste
- Standard fluoride (Experimental): Participants in this arm used standard fluoride containing toothpaste twice daily for routine oral hygiene during the study period.
  Interventions: Other: Standard fluoride toothpaste

INTERVENTIONS:
Other: Propolis Containing Toothpaste — Participants were instructed to brush their teeth using propolis toothpaste twice daily (morning and evening) for 14 days as part of their routine oral hygiene.
  Arms: Propolis containing toothpaste
Other: Probiotic containing toothpaste — Participants were instructed to brush their teeth using probiotic toothpaste twice daily (morning and evening) for 14 days as part of their routine oral hygiene.
  Arms: probiotic containing toothpaste
Other: Phosphate-based formulation toothpaste — Participants were instructed to brush their teeth using Phosphate-based formulation toothpaste twice daily (morning and evening) for 14 days as part of their routine oral hygiene.
  Arms: Phosphate-based formulation toothpaste
Other: Standard fluoride toothpaste — Participants were instructed to brush their teeth using standard fluoride toothpaste twice daily (morning and evening) for 14 days as part of their routine oral hygiene.
  Arms: Standard fluoride

SUMMARY:
This study aimed to evaluate the effects of different toothpaste formulations on oral malodor in young adults, addressing the lack of clinical evidence regarding propolis- and probiotic-containing toothpastes, which have predominantly been investigated in mouthrinse, tablet, or chewing gum formulations.

Volunteers aged 18-30 years with baseline organoleptic assessment (OA) and Breath Checker® (BC) scores >0 were randomized into four toothpaste groups: propolis-containing (Glimo Beta), probiotic-containing (Glimo Pi), phosphate-based (Glimo Gamma), and a standard fluoride toothpaste (Sensodyne). Allocation concealment was ensured using identical coded containers, and outcome assessors were blinded. After exclusions, 52 participants completed the study. Oral malodor was evaluated at baseline (T0) and Day 14 (T1) using OA, BC measurements, and self-perceived oral malodor scores.

ELIGIBILITY:
Inclusion Criteria:

* • No systemic diseases or medications known to cause halitosis

  * No active periodontal disease requiring treatment
  * No antibiotic use within the previous month
  * No orthodontic or removable space-maintaining appliances
  * Non-smokers
  * Organoleptic score >0 and Breath-Checker® (BC) score >0 at baseline

Exclusion Criteria:

* Participants reporting systemic conditions, active periodontal therapy, smoking, or antibiotic usage were excluded.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Change in oral malodor severity | Baseline and Day 14
  Oral malodor was assessed using an organoleptic scoring method and a portable breath checker device. The change in scores from baseline to the end of the intervention period was evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Cankiri Karatekin University, Çankırı, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly due to privacy and ethical considerations.